CLINICAL TRIAL: NCT04046549
Title: A Phase 2a Single-arm, Prospective, Open-label Pilot Study to Evaluate the Safety and Efficacy of Dual Costimulation Blockade With VIB4920 and Belatacept for Prophylaxis of Allograft Rejection in Adults Receiving a Kidney Transplant
Brief Title: A Study to Evaluate the Safety and Efficacy of Dual Costimulation Blockade With VIB4920 and Belatacept for Prophylaxis of Allograft Rejection in Adults Receiving a Kidney Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VIB4920.P2.S1
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Allografts; Rejection; Transplant, Kidney; Transplant Rejection; Kidney Transplantation
Keywords: Renal allograft dysfunction; Cell-mediated rejection; Antibody mediated rejection; Immunosuppression; Acute rejection; VIB4920; MEDI4920; Belatacept; Thymoglobulin; Methylprednisolone; Corticosteroids
MeSH Terms: conditions — Rejection, Psychology | interventions — Abatacept; thymoglobulin; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belatacept+VIB4920 (Experimental): Participants will be admitted to the transplant center for the administration of VIB4920 and belatacept (with Thymoglobulin and corticosteroids) and will be discharged on Day 3/4 at the discretion of the investigator. Participants will return to the study center to receive study drugs (VIB4920 and /or belatacept) weekly for 2 visits, then every 2 weeks for 5 visits, and then monthly for 9 visits for safety monitoring.
  Interventions: Drug: Belatacept; Drug: VIB4920; Drug: Thymoglobulin; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Belatacept — Protocol versions 1 through 4: Belatacept 10 mg/kg by intravenous (IV) infusion on post-op Day 1, repeated on post-op Day 3 or 4 (timing is at investigator's discretion), and at the end of Weeks 2, 4, 8 and 12; then 5 mg/kg IV every 4 weeks from Week 16 to Week 48.
Drug: VIB4920 — Protocol versions 1 and 2: VIB4920 1500 mg by IV infusion on post-op Days 1 and 14, and at the end of Weeks 4, 6, 8 and 10; then 1500 mg every 4 weeks from Week 12 to Week 48.
  Protocol versions 3 and 4: VIB4920 1500 mg by IV infusion on post-op Days 1, repeated on post-op Day 3 or 4 (timing is at investigator's discretion), Week 2, and at the end of Weeks 4, 6, 8, and 10; then 1500 mg every 4 weeks from Week 12 to Week 48.
Drug: Thymoglobulin — Protocol versions 1 and 2: Thymoglobulin 3.0 mg/kg by intravenous (IV) infusion prior to reperfusion of the allograft on the day of transplantation surgery (Day 0) (1 dose).
  Protocol versions 3 and 4: Thymoglobulin 1.5 mg/kg by intravenous infusion prior to reperfusion of the allograft on the day of transplantation surgery (Day 0), prior to VIB4920+belatacept infusion on post-op Day 1, on post-op Day 2, and prior to VIB4920+belatacept infusion on post-op Day 3 or 4.
Drug: Methylprednisolone — Protocol versions 1 and 2: Methylprednisolone by IV infusion (500, 250, 125 and 60 mg on Days 0, 1, 2 and 3, respectively) followed by oral administration of prednisone 30 mg per day on Days 4, 5, and 6.
  Protocol versions 3 and 4: Methylprednisolone by IV infusion (500, 250, 125 and 60 mg on Days 0, 1, 2 and 3, respectively) followed by oral administration of prednisone 30 mg per day on Days 4, 5, 6 and 7. Participants may be tapered to at least 20 mg per day on Day 8, to at least 10 mg per day on Day 15, and to at least 5 mg per day on Day 22. Discontinuation of prednisone following the post-op Day 28 visit.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of dual costimulation blockade with VIB4920 in combination of belatacept in adult male or female recipients of a renal allograft from a deceased, living unrelated or human leukocyte antigen (HLA) non-identical living related donor.

DETAILED DESCRIPTION:
Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a first renal transplant from standard criteria deceased, living unrelated or HLA non-identical living related donor.
* Recipients who are at low immunologic risk:

  1. No donor specific antibodies (DSA), and
  2. Negative cross-match testing.
* Recipients with up to date vaccination as per local immunization schedules.
* Male and female participants who agree to follow protocol defined contraceptive methods.

Exclusion Criteria:

* Participants receiving an allograft from an ABO-incompatible donor.
* Participants treated with systemic immunosuppressive drug therapy for more than a total of 2 weeks within 24 weeks prior to informed consent form signature.
* Participants who have undergone lymphodepleting therapy.
* Participants with medical history of confirmed venous thromboembolism, arterial thrombosis, coagulopathy or known platelet disorders.
* Participants with risk factors for venous thromboembolism or arterial thrombosis, prothrombotic status.
* Participants requiring treatment with antithrombotic drugs (clopidogrel, prasugrel, warfarin, others).
* Participants requiring long-term systemic anticoagulation after transplantation, which would interfere with obtaining biopsies.
* Participants with any contraindication to kidney biopsy.
* Cytomegalovirus (CMV)-seronegative recipients of a CMV-seropositive donor kidney, or unknown CMV serostatus.
* Epstein-Barr virus (EBV)-seronegative or with unknown EBV serostatus.
* Receipt of live (attenuated) vaccine within the 4 weeks before screening.
* Participants with high potential of graft loss due to recurrence of underlying kidney disease.
* Prior solid organ transplant or potential to require a concurrent organ or cell transplant.
* Previous treatment with belatacept and cluster of differentiation 40 (CD40) or anti-CD40L agents.
* Use of B cell depleting therapy, non-depleting B cell directed therapy e.g., belimumab or abatacept within 1 year prior to enrolment.
* At screening blood tests any of the following:

  1. Aspartate aminotransferase (AST) > 2.5 × upper limit of normal (ULN)
  2. Alanine aminotransferase (ALT) > 2.5 × ULN
  3. Alkaline phosphatase (ALP) > 2.5 × ULN
  4. Total bilirubin (TBL) > 2 × ULN
  5. Hemoglobin < 75 g/L
  6. Neutrophils < 1.5 × 10^9/L
  7. Platelets < 100 × 10^9/L
* Participants with severe systemic infections, current or within the 2 weeks prior to transplant surgery.
* Positive test for chronic hepatitis B infection at screening or within the last 12 months.
* Positive test for hepatitis C virus antibody at screening or within the last 12 months.
* Positive test for human immunodeficiency viruses antibody at screening or within the last 12 months.
* History of or active tuberculosis (TB), or a positive QuantiFERON®-TB Gold test at screening, unless previously treated for latent tuberculosis.
* History of cancer, except as follows:

  1. In situ carcinoma of the cervix treated with apparent success with curative therapy > 12 months prior to screening; or
  2. Cutaneous basal cell or squamous cell carcinoma treated with apparent success with curative therapy.
* Lactating or pregnant females.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2023-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - Keck Medical Center of USC, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Duke University School of Medicine, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 25 participants underwent transplant surgery (enrolled); two of these participants were not treated, and are not included in any analysis. A total of 3 participants were enrolled prior to protocol version 3.
Groups:
- Belatacept+VIB4920: Belatacept (protocol versions [v]1-4): 10 mg/kg by intravenous (IV) infusion on post-op Day 1, repeated on post-op Day 3 or 4, and at the end of Weeks 2, 4, 8, 12; then 5 mg/kg IV every 4 weeks from Week 16 to Week 48.
  VIB4920 (protocol v1-2): 1500 mg by IV infusion on post-op Days 1 and 14, and at the end of Weeks 4, 6, 8, 10; then 1500 mg every 4 weeks from Week 12 to Week 48. Protocol v3-4: 1500 mg by IV infusion on post-op Days 1, repeated on post-op Day 3 or 4, Week 2, and at the end of Weeks 4, 6, 8, 10; then 1500 mg every 4 weeks from Week 12 to Week 48.
  Thymoglobulin (protocol v1-2): 3.0 mg/kg by IV infusion prior to reperfusion of the allograft on the day of transplantation surgery (Day 0). Protocol v3-4: 1.5 mg/kg by IV infusion prior to reperfusion of the allograft on the day of transplantation surgery (Day 0), prior to VIB4920+belatacept infusion on post-op Day 1, on post-op Day 2, and prior to VIB4920+belatacept infusion on post-op Day 3 or 4.
  Methylprednisolone (protocol v1-2): IV infusion (500, 250, 125, 60 mg on Days 0, 1, 2, 3, respectively); oral administration of prednisone 30 mg per day on Days 4, 5, 6. Protocol v3-4: IV infusion (500, 250, 125, 60 mg on Days 0, 1, 2, 3, respectively); oral administration of prednisone 30 mg per day on Days 4, 5, 6 and 7. Participants may be tapered to ≤ 20 mg per day on Day 8, to ≤ 10 mg per day on Day 15, and to ≤ 5 mg per day on Day 22. Discontinuation of prednisone following the post-op Day 28 visit.
Period: Overall Study
Arm/Group | Belatacept+VIB4920
Started (enrolled and treated) | 23
Enrolled Prior to Protocol V3.0 | 3
Completed | 13
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3
Not completed — Other, Not Specified | 5

BASELINE CHARACTERISTICS:
Arm/Group | Belatacept+VIB4920
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treated Biopsy-proven Acute Rejection (tBPAR) of Grade 1A or Higher, Graft Loss or Death at Week 24
Description: Histological grading of acute allograft rejection from biopsy specimens was based on Banff criteria 2017. Grade IA: Moderate tubulitis and at least moderate total cortical inflammation and at least moderate scarred cortical inflammation and other known causes ruled out. Grade IB: Severe tubulitis and at least moderate total cortical inflammation and at least moderate scarred cortical inflammation and other known causes ruled out. Grade II. Arterial intimal fibrosis with mononuclear cell inflammation, formation of neointima.
Time Frame: Week 24
Population: Efficacy Evaluable Set: All participants who received the revised regimen of Thymoglobulin and steroids, and any dose of investigational product (IP). Participants enrolled in protocol v3 - 4 were included in the analysis.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Belatacept+VIB4920: Belatacept (protocol versions [v]3-4): 10 mg/kg by intravenous (IV) infusion on post-op Day 1, repeated on post-op Day 3 or 4, and at the end of Weeks 2, 4, 8, 12; then 5 mg/kg IV every 4 weeks from Week 16 to Week 48.
  VIB4920 (protocol v3-4): 1500 mg by IV infusion on post-op Days 1, repeated on post-op Day 3 or 4, Week 2, and at the end of Weeks 4, 6, 8, 10; then 1500 mg every 4 weeks from Week 12 to Week 48.
  Thymoglobulin (protocol v3-4): 1.5 mg/kg by IV infusion prior to reperfusion of the allograft on the day of transplantation surgery (Day 0), prior to VIB4920+belatacept infusion on post-op Day 1, on post-op Day 2, and prior to VIB4920+belatacept infusion on post-op Day 3 or 4.
  Methylprednisolone (protocol v3-4): IV infusion (500, 250, 125, 60 mg on Days 0, 1, 2, 3, respectively); oral administration of prednisone 30 mg per day on Days 4, 5, 6 and 7. Participants may be tapered to ≤ 20 mg per day on Day 8, to ≤ 10 mg per day on Day 15, and to ≤ 5 mg per day on Day 22. Discontinuation of prednisone following the post-op Day 28 visit.
Arm/Group | Belatacept+VIB4920
Number analyzed (Participants) | 20
percentage of participants | 25.0 [12.7 to 41.5]

2. Secondary Outcome: Percentage of Participants With Treated Biopsy-proven Acute Rejection (tBPAR) of Grade 1A or Higher, Graft Loss or Death at Weeks 12 and 48
Description: as for outcome 1
Time Frame: Weeks 12 and 48
Population: Efficacy Evaluable Set: All participants who received the revised regimen of Thymoglobulin and steroids, and any dose of IP. Participants enrolled in protocol v3 - 4 were included in the analysis.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Belatacept+VIB4920: Belatacept (protocol versions [v]3-4): 10 mg/kg by IV infusion on post-op Day 1, repeated on post-op Day 3 or 4, and at the end of Weeks 2, 4, 8, 12; then 5 mg/kg IV every 4 weeks from Week 16 to Week 48.
  VIB4920 (protocol v3-4): 1500 mg by IV infusion on post-op Days 1, repeated on post-op Day 3 or 4, Week 2, and at the end of Weeks 4, 6, 8, 10; then 1500 mg every 4 weeks from Week 12 to Week 48.
  Thymoglobulin (protocol v3-4): 1.5 mg/kg by IV infusion prior to reperfusion of the allograft on the day of transplantation surgery (Day 0), prior to VIB4920+belatacept infusion on post-op Day 1, on post-op Day 2, and prior to VIB4920+belatacept infusion on post-op Day 3 or 4.
  Methylprednisolone (protocol v3-4): IV infusion (500, 250, 125, 60 mg on Days 0, 1, 2, 3, respectively); oral administration of prednisone 30 mg per day on Days 4, 5, 6 and 7. Participants may be tapered to ≤ 20 mg per day on Day 8, to ≤ 10 mg per day on Day 15, and to ≤ 5 mg per day on Day 22. Discontinuation of prednisone following the post-op Day 28 visit.
Arm/Group | Belatacept+VIB4920
Number analyzed (Participants) | 20
percentage of participants
  Week 12 | 25.0 [12.7 to 41.5]
  Week 48 | 25.0 [12.7 to 41.5]

3. Secondary Outcome: Percentage of Participants With Treated Biopsy-proven Acute Rejection (tBPAR), Graft Loss, Death or Loss to Follow-up (LTFU)
Description: as for outcome 1
Time Frame: Week 12, 24, 48
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept+VIB4920
Number analyzed (Participants) | 20
percentage of participants
  Week 12 | 25.0 [12.7 to 41.5]
  Week 24 | 25.0 [12.7 to 41.5]
  Week 48 | 25.0 [12.7 to 41.5]

4. Secondary Outcome: Percentage of Participants With Antibody-Mediated Rejection
Description: The diagnosis of antibody-mediated rejection was based on Banff criteria 2017 - a set of standardized guidelines used by pathologists and clinicians to diagnose and classify rejection based on specific features observed in biopsy samples from the transplanted organ, such as the presence of certain types of immune cells, inflammation, and injury patterns.
Time Frame: Week 12, 24, 48
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept+VIB4920
Number analyzed (Participants) | 20
percentage of participants
  Week 12 | 10.0 [2.7 to 24.5]
  Week 24 | 10.0 [2.7 to 24.5]
  Week 48 | 15.0 [5.6 to 30.4]

5. Secondary Outcome: Percentage of Participants With Treated Biopsy-proven Acute Rejection (tBPAR)
Description: Histological grading of acute allograft rejection from biopsy specimens was based on Banff criteria 2017. Grade IA: Moderate tubulitis and at least moderate total cortical inflammation and at least moderate scarred cortical inflammation and other known causes ruled out. Grade IB: Severe tubulitis and at least moderate total cortical inflammation and at least moderate scarred cortical inflammation and other known causes ruled out. Grade II. Arterial intimal fibrosis with mononuclear cell inflammation, formation of neointima. tBPAR was defined as a BPAR which was treated with anti-rejection therapy.
Time Frame: Week 12, 24, 48
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept+VIB4920
Number analyzed (Participants) | 20
percentage of participants
  Week 12 | 25.0 [12.7 to 41.5]
  Week 24 | 25.0 [12.7 to 41.5]
  Week 48 | 25.0 [12.7 to 41.5]

6. Secondary Outcome: Percentage of Participants With Biopsy Proven Acute Rejection (BPAR)
Description: as for outcome 1
Time Frame: Week 12, 24, 48
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept+VIB4920
Number analyzed (Participants) | 20
percentage of participants
  Week 12 | 25.0 [12.7 to 41.5]
  Week 24 | 25.0 [12.7 to 41.5]
  Week 48 | 25.0 [12.7 to 41.5]

7. Secondary Outcome: Percentage of Participants With Treated Acute Rejections
Description: Acute rejections, per clinical judgement of the investigator followed by confirmatory biopsy, were treated with bolus methylprednisolone (other corticosteroids were acceptable at an equivalent dose) according to local practice.
Time Frame: Week 12, 24, 48
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept+VIB4920
Number analyzed (Participants) | 20
percentage of participants
  Week 12 | 25.0 [12.7 to 41.5]
  Week 24 | 25.0 [12.7 to 41.5]
  Week 48 | 30.0 [16.7 to 46.7]

8. Secondary Outcome: Percentage of Participants With De Novo Donor-specific Antibodies (dnDSA)
Description: Serum samples were collected for de novo donor-specific antibodies (dnDSA) using solid phase (bead-based) assays.
Time Frame: Week 12, 24, 48
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From written informed consent signature (Day -28 to -1) and the end of the safety follow-up 60 weeks (up to 64 weeks) Adverse Events: From first dose of study drug until the end of treatment + 12 weeks (up to 60 weeks)
Description: As it is in our pre-specified analysis, all safety data was based on safety analysis set, i.e., all subjects who received any dose of IP.
Arm/Group | Belatacept+VIB4920
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 10/23
Other Adverse Events (participants affected / at risk) | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept+VIB4920 (N=23)
Ileus (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Kidney transplant rejection (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | 2
Blood creatinine increased (Investigations) | 1
Cytomegalovirus test positive (Investigations) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Depression suicidal (Psychiatric disorders) | 1
Subcapsular renal haematoma (Renal and urinary disorders) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept+VIB4920 (N=23)
Anaemia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 2
BK virus infection (Infections and infestations) | 4
COVID-19 (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 2
Procedural pain (Injury, poisoning and procedural complications) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04046549/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT04046549/SAP_001.pdf